CLINICAL TRIAL: NCT01944904
Title: Study of the Effect of Prebiotic Xylooligosaccharide (XOS) on Microbita and Blood Glucose
Brief Title: Investigation of the Ability of a Supplement to Increase Good Bacteria in the Human Intestine and Blood Sugar Levels
Acronym: XOS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XOS2 053113
Record Dates: First submitted 2013-09-04; First posted 2013-09-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Pre-diabetic
Keywords: XOS; pre-diabetic; abnormal glucose levels
MeSH Terms: conditions — Glucose Intolerance | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Subjects will be asked to take the dietary supplement daily for 8 weeks. Blood samples will be taken at screen, baseline and week 8. An oral glucose tolerance test will be taken at baseline and week 8. Additionally subjects will be asked to collect their stool samples at Baseline, week 4, and 8. Subjects will also undergo a test to determine their body composition at baseline and week 8. Subjects will be asked to keep a diary of their bowel habits and any symptoms that might be related to the supplement. Subjects will be asked to recall the foods that they have eaten in the past 24 hours and to avoid any foods that contain XOS and probiotic bacteria during the study.
  Interventions: Dietary Supplement: Sugar Pill
- XOS 2.8 (Active Comparator): Subjects will be asked to take the dietary supplement daily for 8 weeks. Blood samples will be taken at screen, baseline and week 8. An oral glucose tolerance test will be taken at baseline and week 8. Additionally subjects will be asked to collect their stool samples at Baseline, week 4, and 8. Subjects will also undergo a test to determine their body composition at baseline and week 8. Subjects will be asked to keep a diary of their bowel habits and any symptoms that might be related to the supplement. Subjects will be asked to recall the foods that they have eaten in the past 24 hours and to avoid any foods that contain XOS and probiotic bacteria during the study.
  Interventions: Dietary Supplement: XOS 2.8

INTERVENTIONS:
Dietary Supplement: Sugar Pill — The placebo is identical in appearance to the XOS and contains 505mg maltodextrin
  Arms: Sugar Pill
Dietary Supplement: XOS 2.8 — 2.8g XOS is white or off-white crystalline substance and contains 500mg XOS 70P and 20mg maltodextrin
  Arms: XOS 2.8

SUMMARY:
This study aims to determine whether the use of a supplement called xylooligosaccharide (XOS) increases the number of good bacteria that live in human intestines and can maintain healthy blood sugar levels, and whether XOS has any unpleasant or unexpected side effects when consumed at different dosages. Subjects who participate in this study will be randomized to receive an eight week supply of either a lower dose of XOS or placebo (no active substance). This will be determined randomly, in a process similar to flipping a coin. Blood samples will be taken at each visits, including an oral glucose tolerance test. Subjects will also be asked to collect and bring in stool samples at three different time points during the study.

Subjects will have a 50/50 chance of being assigned to the either study group. This is a double-blind study which means neither the study investigator nor the subject will know to which group he/she has been assigned. In case of an emergency, the study doctor can get this information.

DETAILED DESCRIPTION:
Prebiotics are highly effective and important for many applications in medicine. They are not absorbed and do not contribute to human nourishment, but rather exert a profound effect on the human bowel flora. The principal effect on the human bowel flora is to stimulate the growth of Bifidobacterium and Lactobacillus species. These are benign organisms in that they are seldom involved in infections or other pathological processes. However, numerous health promoting benefits of these bacterial genera have been noted, with effects on infectious and non-infectious disease. They induce host genes involved in innate immunity, sometimes in collaboration with other elements of the gut flora such as Bacteroides thetaiotaomicron and Lactobacillus casei. Animal studies 2 indicate a protective effect against bacterial translocation from the GI tract. An extensive cataloguing of genomes of bifidobacteria and other intestinal bacteria reveals that the bifids play a very significant role in many important areas such as carbohydrate, amino acid, nucleotide, lipid, inorganic ion transport and metabolism; energy production and conversion; cell wall and membrane biogenesis; signal transduction mechanisms; transcription and translation; and defense mechanisms .

The metabolic syndrome which includes non-alcoholic fatty liver disease, obesity, and insulin resistance has responded to prebiotics in rodent trials; it is estimated that 20-30% of populations in developed countries have this disease. Parnell and Reimer have demonstrated that prebiotics oligofructose supplementation has the potential to promote weight loss and improve glucose regulation in overweight adults likely through suppressed ghrelin and enhanced PYY1.

The investigators have completed a study at UCLA studying the effects of XOS on human microbiota. There were three phases including a 2-week run-in period, 8-week intervention period, and a 2-week washout. Thirty two volunteers were randomly assigned to take a supplement containing 1.4 g XOS (1.4g XOS 70P), 2.8 g XOS (2.8g XOS 70P) or placebo.

Total of 32 subjects were enrolled into the study. One subject from the placebo group and one from the low dose group dropped out of the study for non specific gastrointestinal complaint.

Altogether, 120 stool samples were received from 11 low dose subjects, 9 high dose subjects, and 10 placebo group subjects. Bacterial culture was performed from all the 120 stool samples received. One placebo group subject, two high dose group subjects, and two low dose group subjects were excluded from the analyses because of compromised specimen quality.

The Bifidobacterium counts of the subjects after high dose XOS intervention was significantly higher from the base line at 4, 8, and 10 weeks. Similarly, the increase of Bifidobacterium counts was significantly higher in the high XOS group at 4 weeks compared to the low XOS group. The low XOS group had significantly higher Bifidobacterium counts compared to the placebo group subjects at 8 and 10 weeks. The total anaerobic flora counts and to some degree the total aerobic flora counts of the subjects after high dose XOS intervention were significantly higher from the base-line at 4 and 8 weeks. The mean changes of total anaerobic flora counts were significantly higher in the high XOS group at 4, 8, and 10 weeks compared to the placebo group. Interestingly, also Bacteroides fragilis group counts of the subjects after high dose XOS intervention were significantly higher from the base line at 4, 8, and 10 weeks and the mean changes were significantly higher in the high XOS group compared to the low and placebo groups. There were no major significant differences in the counts of Lactobacillus sp., Enterobacteriaceae, and clostridia between the three dose groups evaluated

The XOS was tolerated well by all study subjects (normal adult). At base-line, most of the subjects had relatively high counts of Bifidobacterium species with lower counts of Lactobacillus species. Several different species of each of these genera were present. Bifidobacterium species showed significant increases in counts in subjects on XOS supplementation, with the higher dose group showing significantly greater increases than the lower dose group. Both high and low dose groups showed significantly higher counts of Bifidobacterium sub-species than the placebo group. Lactobacillus species counts did not increase significantly in subjects on XOS supplementation. There was a statistically significant increase in the counts of the B. fragilis group at all time periods for the high dose XOS group. As mentioned before, bifidobacteria may induce host genes involved in innate immunity in collaboration with other elements of the gut flora such as B. fragilis group. The increase in the counts of the "total anaerobes" reflects the increased counts in the Bifidobacterium and B. fragilis group, both of which are anaerobic. Some Bifidobacterium species may grow aerobically as well, which may be reflected in the modest increase of the aerobic counts in the high dose XOS group. In this study, the XOS supplementation had no significant effect on stool pH or SCFAs.

The investigators propose to conduct a 10 week, randomized, placebo controlled, two arm study with 20 subjects with metabolic syndrome. Subjects will be randomly assigned to take a powder mixture containing 2.8 g XOS (2.94g XOS 95P) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-70 years of age at screen
2. BMI between 27 to 35
3. Fasting glucose level >100 mg/dL or >200 mg/dL at 1 hour after ingesting of 75 grams of glucose
4. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent

Exclusion Criteria:

1. Any subject with a history of diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
2. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
3. Any subject who currently uses tobacco products.
4. Any history of gastrointestinal disease except for appendectomy
5. No antibiotics or laxatives use during the 2 months before the study.
6. Any subject who is unable or unwilling to comply with the study protocol.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The Effects of Xyloologosarcharide (XOS) on colonic flora in volunteers with abnormal glucose levels | 10 weeks
  After 2 weeks of run-in, 20 healthy volunteers with fasting glucose level >100 mg/dL or >200 mg/dL at 1 hour after ingesting of 75 grams of glucose will be randomly assigned to take 2.8 grams/day or placebo for 8 weeks. The bifidobarteria counts will be assessed at screening, baseline and 8 weeks on supplementation of XOS and cessation of XOS.

SECONDARY OUTCOMES:
The Effects of Xyloologosarcharide (XOS) on glucose and insulin | 10 weeks
  Glucose, insulin and triglyceride levels will be tested at time 0, 30 min, 60 min, and 120 min after 75 grams of glucose load at baseline and 8 weeks.

OTHER OUTCOMES:
The effects of Xylooligosaccharide (XOS) on body weight and body composition | 10 weeks
  Body weight and body composition will be measured at baseline and week 8.

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, PhD, Principal Investigator — University of California, Los Angeles; Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Result] Yang J, Summanen PH, Henning SM, Hsu M, Lam H, Huang J, Tseng CH, Dowd SE, Finegold SM, Heber D, Li Z. Xylooligosaccharide supplementation alters gut bacteria in both healthy and prediabetic adults: a pilot study. Front Physiol. 2015 Aug 7;6:216. doi: 10.3389/fphys.2015.00216. eCollection 2015. PMID 26300782